CLINICAL TRIAL: NCT05284136
Title: Prospective rAndomized Controlled tRial of Crohn's diseAse Exclusion Diet vs corticosteroIds in patientS With activE Crohn's Disease - PARADISE
Brief Title: Exclusion Diet vs corticosteroIds in patientS With activE Crohn's Disease
Acronym: PARADISE
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP200030
Record Dates: First submitted 2022-02-28; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-02

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Diet; Corticosteroids
MeSH Terms: conditions — Crohn Disease | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crohn's disease exclusion diet (CDED) (Experimental): 16-week course of Crohn's disease exclusion diet (CDED) and Partial Enteral Nutrition.
  Interventions: Dietary Supplement: Crohn's disease exclusion diet (CDED)
- Steroids (Active Comparator): oral prednisolone at an initial dose of 40 to 60 mg/day.
  Interventions: Drug: Oral prednisolone

INTERVENTIONS:
Dietary Supplement: Crohn's disease exclusion diet (CDED) — 16-week course of CDED+Partial Enteral Nutrition. During the first 6 weeks (phase 1 of CDED), patients will be prescribed the CDED and oral Modulen 1 liter (1000kcal) daily. Between week 6 and 16 (phase 2 of CDED), patients will be prescribed CDED and oral Modulen (500 mL).
  Arms: Crohn's disease exclusion diet (CDED)
Drug: Oral prednisolone — oral prednisolone at an initial dose of 40 to 60 mg/day (or 1 mg/kg for those patients who weigh less than 40 kg), with a fixed, tapering regimen such that patients should be off steroids by the last day of week 12. Increases in steroid dose during tapering of corticosteroids is allowed but if the patient receives steroids (other than hydrocortisone for adrenal insufficiency) after week 12, he/she is in failure.
  Arms: Steroids

SUMMARY:
Crohn's disease exclusion diet (CDED) is a whole-food diet coupled with partial enteral nutrition. The main objective of this trial is to assess whether CDED is superior to corticosteroids, in terms of endoscopic response, in patients active CD. The primary endpoint is endoscopic response at week 16, without corticosteroids or further therapeutic intervention, assessed by a centralized, anonymous and blinded, double lecture panel of panenteric PillCam Crohn's Capsule. This is a multicentre, open-label, comparative, randomized, 2:1, controlled, single-blind, superiority trial. Patients included are aged 16 to 70 years, have mild to moderate, luminal, active CD, and have active endoscopic lesions. Eighty patients will be randomized between CDED (n=56) and corticosteroids (n=24) in centres in France, Israel and the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 to 70 years,
* With mild to moderate, luminal, active CD, defined by a CDAI of 150 to 350,
* Involving the small bowel, and/or the colon
* Not treated with corticosteroids at baseline
* Patent small bowel as assessed by the patency capsule
* Active endoscopic lesions, as defined by Lewis score ≥ 225 in the small bowel and/or SES-CD≥ 4 in the colon. The eligibility of the patient will be determined by the site investigator and a central reader.
* Informed consent to participate in this study. In patients from France and Israel who are aged less than 18: parents' informed consent to participate in this study (parents' agreement is not required in patients aged 16 to 18 in the Netherlands)
* Affiliation to social security or any health insurance

Exclusion Criteria:

* Inability to follow the CDED during 16 weeks.
* Prior intolerance to corticosteroids.
* Ongoing infections, evolving virus diseases.
* Live vaccines.
* Psychotic state not controlled by treatment.
* Arthritis or uveitis as main presenting symptoms.
* Patients with severe and/or predominant rectal or perianal disease.
* Heavy smokers (more than 10 cigarettes per day).
* Infliximab, adalimumab, methotrexate or azathioprine initiated less than 3 months before inclusion in this trial.
* Vedolizumab, ustekinumab initiated less than 6 months before inclusion in this trial.
* Change in methotrexate, azathioprine, infliximab, adalimumab, vedolizumab or ustekinumab dosage less than 3 months before inclusion.
* Pregnant or lactating women.
* Patients already included in a biomedical research other than an observational study (e.g. registry, cohort, biobank).
* Severe pubertal delay (Tanner 1 or Tanner 2) and/or height velocity z-score < 2.5 and/or Bone mineral density z-score (hip or lumbar spine) <2.5.
* Persons deprived of their liberty by a judicial or administrative decision, persons subject to psychiatric care under sections L.3212-1 et L.3213-1 and persons admitted to a health or social institution for purposes other than research (L.1121-6)

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Endoscopic response W16 | Week 16
  The primary endpoint is the endoscopic response at week 16, assessed by Panenteric capsule (PillCam Crohn's capsule) using centralized, anonymous and blinded reading of PCC. The response is defined as a single binary endpoint according to the initial strata of the patient:
  * Small bowel Crohn's diseAse (CD) : decrease of the Lewis score of at least 50% compared to baseline values
  * Colonic CD : decrease of SES-CD of at least 50% compared to baseline values
  * Small bowel and colonic CD : decrease of the Lewis score of at least 50% AND decrease of SES-CD of at least 50% compared to baseline values.
  Lewis score : Gralnek IM, Defranchis R, et al. Development of a capsule endoscopy scoring index for small bowel mucosal inflammatory change. Aliment Pharmacol Ther 2008; 27: 146-154.
  SES-CD : Daperno M, D'Haens G, et al . Development and validation of a new, simplified endoscopic activity score for Crohn's disease: the SES-CD. Gastrointest Endosc 2004; 60 (4): 505-512.

SECONDARY OUTCOMES:
Rate of Clinical remission | Week 16 and Week 48
  Crohn's disease activity index (CDAI) <150. CDAI will be measured by the investigator on the basis of prospective questionnaires filled in by patients during the week preceding each visit.
  Best, William R., Jack M. Becktel, John W. Singleton, and Fred Kern Jr. "Development of a Crohn's disease activity index: National Cooperative Crohn's Disease Study." Gastroenterology 70, no. 3 (1976): 439-444.
Rate of Clinical response | Week 16 and Week 48
  Decrease of at least 70 points in Crohn's disease activity index (CDAI) compare to CDAI baseline.
Rate of Need for further therapeutic intervention | Week 48
  Need for further therapeutic intervention (i.e., steroids, immunosuppressants, new biologic or surgery) between week 13 and 48
Decrease of fecal calprotectin concentration | Week 16 and Week 48
  Decrease of fecal calprotectin of at least 50% compared to baseline at week 16 and 48
Rate of Fecal calprotectin below thresholds | Week 16
  Fecal calprotectin of less than 250 μg/g, less than 100 μg/g and less than 50 μg/g at week 16.
Rate of normal CRP concentration | Week 16 and Week 48
  CRP serum level <5 mg/L.
Rate of Endoscopic remission | Week 16
  Endoscopic remission as defined as Lewis score <135 in the small bowel and/or Simple Endoscopic Score for Crohn Disease (SES-CD) <4 in the colon, without further therapeutic intervention (surgery, biologics or dietary intervention) at week 16.
  Dias de Castro, F., Pedro Boal Carvalho, Sara Monteiro, Bruno Rosa, João Firmino-Machado, Maria João Moreira, and José Cotter. "Lewis score-prognostic value in patients with isolated small bowel Crohn's disease." Journal of Crohn's and Colitis 9, no. 12 (2015): 1146-1151.
  Daperno, Marco, Geert D'Haens, Gert Van Assche, Filip Baert, Philippe Bulois, Vincent Maunoury, Raffaello Sostegni et al. "Development and validation of a new, simplified endoscopic activity score for Crohn's disease: the SES-CD." Gastrointestinal endoscopy 60, no. 4 (2004): 505-512.
Rate of Endoscopic response | Week 16
  Endoscopic response and remission graded by Eliakim score at week 16.
  Eliakim, Rami, et al. "A novel PillCam Crohn's capsule score (Eliakim score) for quantification of mucosal inflammation in Crohn's disease." United European gastroenterology journal 8.5 (2020): 544-551.
Gut microbiota composition | Week 6 and Week 16
  Gut microbiota composition at week 6 and week 16. The endpoint consist in the rate of the diffrent microorganisms present in the gut.
Value of adherence by Medication Adherence Report Scale | Week 1, Week 9 and Week 16
  Medication Adherence Report Scale (MARS) at week 1, 9 and 16.
  Chan, Amy Hai Yan, Rob Horne, Matthew Hankins, and Claudia Chisari. "The medication adherence report scale: a measurement tool for eliciting patients' reports of nonadherence." British Journal of Clinical Pharmacology 86, no. 7 (2020): 1281-1288.
Rate of adherence using food diaries | Week 1, Week 9 and Week 16
  Adherence evaluate as binuary outcome evaluated using food diaries at week 1, 9 and 16
Value of Quality of life | Week 3, Week 6 and Week 16
  Quality of life will be assessed by short inflammatory bowel disease questionnaire (IBDQ) at week 3, 6 and 16.
  Irvine, E. J., Q. Zhou, and A. K. Thompson. "The Short Inflammatory Bowel Disease Questionnaire: A Quality of Life Instrument for Community Physicians Managing Inflammatory Bowel Disease." American Journal of Gastroenterology (Springer Nature) 91.8 (1996).
Value Work | Week 6 and Week 16
  Work productivity and activity will be assessed by thework productivity and activity impairment questionnaire (WPAI) at 6 and 16.
  Reilly, Margaret C., Arthur S. Zbrozek, and Ellen M. Dukes. "The validity and reproducibility of a work productivity and activity impairment instrument." Pharmacoeconomics 4.5 (1993): 353-365.

CONTACTS AND LOCATIONS:
Locations (2):
- Gastroenterology department, Le Kremlin-Bicêtre, France
- Department of Gastroenterology & Hepatology (MDL), Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided